CLINICAL TRIAL: NCT00281099
Title: MVP Trial (Managed Ventricular Pacing ("MVP") Versus Backup Ventricular Pacing at a Rate of 40 Beats Per Minute ("VVI 40") Pacing Trial)
Brief Title: Managed Ventricular Pacing ("MVP") Trial
Acronym: MVP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to reach statistical significance toward primary endpoint
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Steve Erickson, Principal Clinical Trial Leader, Medtronic CRDM
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 240
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Results first posted 2010-08-03 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Heart Disease
Keywords: ICD; Pacing; Heart Failure
MeSH Terms: conditions — Heart Diseases; Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VVI 40 pacing (Active Comparator): Backup ventricular pacing (VVI) at 40 beats per minute
  Interventions: Device: ICD (Implantable Cardioverter Defibrillator)
- MVP pacing (Active Comparator): Managed ventricular pacing (MVP) at 60 beats per minute
  Interventions: Device: ICD (Implantable Cardioverter Defibrillator)

INTERVENTIONS:
Device: ICD (Implantable Cardioverter Defibrillator) — VVI 40 vs. MVP
  Other Names: Intrinsic™; EnTrust™

SUMMARY:
The purpose of the study is to compare two device settings (sets of instructions) used by the ICD. The Implantable Cardiac Defibrillator ("ICD") can be set to use one wire (top or bottom of the heart) or two wires (top and bottom). The study will compare how much time either ICD wire is used by the ICD and the status of congestive heart failure.

DETAILED DESCRIPTION:
Recent research supports the hypothesis that reducing the amount of pacing in the lower right chamber of the heart may prevent the progression of congestive heart failure (CHF) in some implantable cardioverter defibrillator (ICD) patients. CHF refers to symptoms (shortness of breath, fatigue, fluid overload) caused by decreased pumping action of the heart muscle. The ICD can be set to use one wire (top or bottom of the heart) or two wires (top and bottom). Both settings allow the heart to beat more naturally using its own electrical signals. Two device settings will be compared. Managed ventricular pacing (MVP) will allow the ICD to use both wires only as necessary. This setting allows the ICD to send electrical signals to the top and bottom chambers of the heart if needed. The other setting, ventricular pacing (VVI) will allow the ICD to operate the bottom chamber of the heart if it is needed.

ELIGIBILITY:
Inclusion Criteria:

* Conventional indication for ICD therapy according to current evidence-based guidelines and in accordance with the corresponding United States Centers for Medicare and Medicaid Services National Coverage Determination for the use of ICDs.
* Prior myocardial infarction ("MI") and an left ventricular ejection fraction ("LVEF") of less than 30%
* Ischemic Dilated Cardiomyopathy (IDCM), New York Heart Association ("NYHA") Class II or II heart failure, and LVEF less than or equal to 35%
* Non-Ischemic Dilated Cardiomyopathy (NIDCM) greater than 3 months, NYHA Class II or II heart failure, and LVEF less than or equal to 35%
* First ICD implant
* Successful implant with a study device with approved labeling

Exclusion Criteria:

* Failure to meet any of the inclusion criteria
* Class I pacing indication
* Chronic atrial fibrillation ("AF") without any documented sinus mechanism for at least 6 months
* Inability or unwillingness to give informed consent
* Life expectancy less than 12 months or a heart transplant anticipated within 6 months
* Inability to successfully comply with study participation and follow up requirements
* Patient involved in another clinical trial that may confound the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1031 (Actual)
Dates: Start 2004-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael O Sweeney, Principal Investigator — Brigham and Women's Hospital
Locations (73):
- United States (50):
  - Anchorage, Alaska
  - Little Rock, Arkansas
  - North Little Rock, Arkansas
  - Brandon, Florida
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Naples, Florida
  - Pensacola, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Detroit, Michigan
  - Lansing, Michigan
  - Marquette, Michigan
  - Petoskey, Michigan
  - Coon Rapids, Minnesota
  - Saint Paul, Minnesota
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Hackensack, New Jersey
  - Newark, New Jersey
  - New Hyde Park, New York
  - New York, New York
  - Gastonia, North Carolina
  - Raleigh, North Carolina
  - Mayfield Hts., Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Taylorville, Utah
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Sankt Pölten, Austria
- Canada (6):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Ottawa, Ontario
  - Montreal, Quebec
  - Ste-Foy, Quebec
- Aarus, Denmark
- France (2):
  - Le Chesnay
  - Lille
- Germany (5):
  - Bad Berka
  - Franfurt Am Main
  - Heidelberg
  - Homburg/Saar
  - Kiel
- Israel (3):
  - Haifa
  - Milano
  - Tel Aviv
- Milan, Italy
- Tromsø, Norway
- Valencia, Spain
- Zurich, Switzerland
- London, United Kingdom

REFERENCES:
- [Derived] Sweeney MO, Ellenbogen KA, Tang AS, Whellan D, Mortensen PT, Giraldi F, Sandler DA, Sherfesee L, Sheldon T; Managed Ventricular Pacing Versus VVI 40 Pacing Trial Investigators. Atrial pacing or ventricular backup-only pacing in implantable cardioverter-defibrillator patients. Heart Rhythm. 2010 Nov;7(11):1552-60. doi: 10.1016/j.hrthm.2010.05.038. Epub 2010 Jun 4. PMID 20685401

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2051 subjects were screened for the study. Of the 2051 subjects screened, 1037 were enrolled in the study. 6 of 1037 subjects later failed to meet other qualifying inclusion criteria and were not randomized and assigned to a study arm.
Groups:
- VVI 40 Pacing: Backup ventricular pacing at a rate of 40 beats per minute
- MVP Pacing: Managed Ventricular Pacing at a rate of 60 beats per minute
Period: Overall Study
Arm/Group | VVI 40 Pacing | MVP Pacing
Started | 513 | 518
Completed | 308 | 296
Not Completed | 205 | 222
Not completed — Death | 46 | 57
Not completed — Lost to Follow-up | 10 | 19
Not completed — Withdrawal by Subject | 65 | 70
Not completed — Physician Decision | 79 | 72
Not completed — Heart Transplant/Device Exit/Changeout | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VVI 40 Pacing | MVP Pacing | Total
Number analyzed (Participants) | 513 | 518 | 1031
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 289 | 284 | 573
  >=65 years | 224 | 234 | 458
Age Continuous [Mean (Standard Deviation); unit: years] | 61.7 (11.7) | 62.6 (12.0) | 62.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 104 | 212
  Male | 405 | 414 | 819
Region of Enrollment [Number; unit: participants]
  France | 3 | 3 | 6
  United States | 390 | 390 | 780
  Canada | 58 | 60 | 118
  Spain | 2 | 3 | 5
  Austria | 1 | 0 | 1
  Denmark | 4 | 3 | 7
  Israel | 14 | 15 | 29
  Germany | 14 | 16 | 30
  United Kingdom | 7 | 7 | 14
  Switzerland | 9 | 9 | 18
  Italy | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality and Heart Failure-related Urgent Care Visits and Heart Failure ("HF") Hospitalizations.
Description: A composite endpoint of all cause mortality and HF hospitalizations or urgent care. (Emergency Department, Urgent Clinic visits, or hospitalizations wiht intravenous medications for HF)
Time Frame: Enrollment to last visit (up to 45 months post-randomization) or death
Population: 1 of 1031 randomized subjects had a history of at least 6 months of chronic atrial fibrillation ("AF"), which was an exclusion criterion. The remaining 1030 randomized subjects met all inclusion criteria and made up the analysis cohort. An intention to treat analysis was performed for this objective.
Measure: Number; unit: events
Groups:
- VVI 40: Backup ventricular pacing at a rate of 40 beats per minute
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
events | 167 | 188
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; This is a multiple events survival analysis, with time to first primary endpoint, time between successive endpoints, and time from last endpoint to last follow-up visit determined for each subject. The null hypothesis is that the mortality/ heart failure ("HF") urgent care/HF hospitalization hazard rate for patients with no Class I pacing indication and MVP is greater than that of similar patients with VVI 40; Test type: Non-Inferiority or Equivalence — A non-inferiority analysis was performed, with the hazard ratio as the parameter of interest and the non-inferiority threshold of 1.21. The one-sided upper confidence bound for the hazard ratio had to be less than 1.21 for the null hypothesis to be rejected. The threshold of 1.21 was derived by using a noninferiority threshold of a 5 percentage point difference in 24 month event-free rates; Andersen-Gill Model — There were 167 events by 90 subjects in the VVI 40 arm, compared to 188 events among 104 subjects in the MVP arm; An Andersen-Gill model was used to account for multiple primary endpoints per subject; Hazard Ratio (HR) = 1.139, 96.3% CI [1.139 to 1.590] — 4 interim analyses were performed & the O'Brien-Fleming alpha-spending function required a 96.3% confidence interval

2. Secondary Outcome: Occurrence of Worsening Heart Failure-related Adverse Events
Description: HF event meeting primary endpoint definition, or adverse events associated with, but not limited to, any of the following: symptoms or physical signs compatible with worsening HF, laboratory evidence of HF, any modification of oral heart failure therapy
Time Frame: Enrollment to last visit (up to 45 months post-randomization)
Population: as for outcome 1
Measure: Number; unit: participants/events
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
participants/events
  Number of Participants with Events | 96 | 108
  Number of Events | 193 | 190
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; This is a multiple events survival analysis, and so the time from randomization to first HF event, time between successive HF events, and time from last HF event to last follow-up visit was determined for each subject. Since non-inferiority analysis is intended to prove that one therapy is equivalent or superior to another therapy, the null hypothesis being tested is that the worsening HF hazard rate for patients with MVP programming is greater than that of patients with VVI 40 programming; Test type: Non-Inferiority or Equivalence — A non-inferiority analysis was performed, with the hazard ratio as the parameter of interest and the non-inferiority threshold of 1.241. The one-sided upper confidence bound for the hazard ratio had to be less than 1.241 for the null hypothesis to be rejected. The threshold of 1.241 was derived by using a non-inferiority threshold of a 5 percentage point difference in 24 month HF event-free rates; Andersen-Gill Model; An Andersen-Gill model was utilized to account for multiple HF events per subject; Hazard Ratio (HR) = 1.029, 95% CI [1.029 to 1.381]

3. Secondary Outcome: Distribution of Patients by NYHA (New York Heart Association) Functional Class Over Time
Description: NYHA Classification at each scheduled Follow-up visit. The scale for this measure is as follows: NYHA I= best, NYHA IV= worst.
Time Frame: Baseline, 12, 24 and 36 month visits
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
participants
  Baseline NYHA I | 140 | 122
  Baseline NYHA II | 271 | 293
  Baseline NYHA III | 93 | 98
  Baseline NYHA IV | 1 | 1
  Baseline NYHA Obtained Outside Window | 7 | 4
  12 Month NYHA I | 139 | 118
  12 Month NYHA II | 242 | 234
  12 Month NYHA III | 46 | 55
  12 Month NYHA IV | 5 | 1
  12 Month NYHA Missing due to Death | 21 | 22
  12 Month NYHA Missing For Other Reasons | 59 | 88
  24 Month NYHA I | 119 | 104
  24 Month NYHA II | 205 | 197
  24 Month NYHA III | 44 | 44
  24 Month NYHA IV | 2 | 4
  24 Month NYHA Missing due to Death | 39 | 40
  24 Month NYHA Missing For Other Reasons | 103 | 129
  36 Month NYHA I | 18 | 23
  36 Month NYHA II | 46 | 42
  36 Month NYHA III | 8 | 7
  36 Month NYHA IV | 1 | 1
  36 Month NYHA Missing due to Death | 46 | 57
  36 Month NYHA Missing For Other Reasons | 393 | 388
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; A model with covariates for time and randomization arm was fit to test the null hypothesis that the risk of worsening NYHA status over time among patients with MVP programming was equal to that of patients with VVI 40 programming. This analysis combined NYHA IV and Death into one category. The model included interaction terms for time and randomization arm; Test type: Superiority or Other; p > 0.05, Cumulative Logits Model — The a priori alpha level for each covariate was 0.05. The p-value outcome provided is for the randomization arm main effect and all interactions between randomization arm and time; The analysis included data for all four time points (baseline, 12, 24, and 36 months) and all NYHA levels
Statistical Analysis 2: Comparison: VVI 40 vs MVP Pacing; The null hypothesis for this analysis was the same as for the prior analysis: that the risk of worsening NYHA status over time among patients with MVP programming was equal to that of patients with VVI 40 programming. In this analysis, however, death was considered a 5th category in addition to NYHA I-IV. An interaction term for time and randomization arm was also included; Test type: Superiority or Other; p > 0.05, Cumulative Logit Model — The a priori alpha level for each covariate was 0.05. The p-value outcome provided is for the randomization arm main effect and all interaction terms between randomization arm and time; The analysis included data for all four time points (baseline, 12, 24, and 36 months) and all NYHA levels

4. Secondary Outcome: Heart Chamber Dimensions and Wall Thicknesses
Description: Echocardiogram measures for each endpoint were obtained at multiple time points.
Time Frame: Baseline, 12, and 24 month visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
centimeters (cm)
  LV End Diastolic Dimension(LVEDD) (cm) at Baseline | 5.9 (1) | 6 (0.9)
  LVEDD (cm) at 12 Months | 6 (0.9) | 6 (0.9)
  LVEDD (cm) at 24 Months | 6 (1) | 5.9 (0.8)
  LV End Systolic Dimension (LVESD) (cm) at Baseline | 4.9 (1.1) | 4.9 (1)
  LVESD (cm) at 12 Months | 4.7 (1.1) | 4.9 (1)
  LVESD (cm) at 24 Months | 4.8 (1.1) | 4.8 (1.1)
  Septal Thickness (cm) at Baseline | 1 (0.3) | 1 (0.3)
  Septal Thickness (cm) at 12 Months | 1 (0.3) | 1 (0.3)
  Septal Thickness (cm) at 24 Months | 1 (0.3) | 1 (0.2)
  Posterior Wall Thickness (cm) at Baseline | 1 (0.2) | 1 (0.2)
  Posterior Wall Thickness (cm) at 12 Months | 1 (0.2) | 1 (0.2)
  Posterior Wall Thickness (cm) at 24 Months | 1 (0.2) | 1 (0.2)
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; A linear mixed model was fit for each of the followoing: LVEDD, LVESD, Septal Wall Thickness, and Posterior Wall Thickness; the purpose was to test whether patients with MVP and no pacing indication over time had a different average value for that measure than patients with VVI and no pacing indication. Data were also collected from the 36 month visits but were excluded due to the trial being stopped early and only a subset of patients having data for those visits; Test type: Superiority or Other; p > 0.10, Mixed Models Analysis — In each case the a priori threshold for significance for Arm was 0.05; Model fit with time and arm as covariates, the interaction between them included. Interaction shown to not be significant and model refit without it

5. Secondary Outcome: Left Ventricular (LV) Ejection Fraction and Fractional Shortening
Description: Echocardiogram measures for each endpoint were obtained at multiple time points.
  LV Ejection Fraction is the percentage of a patient's blood moved out of the left venricle when the heart pumps. The measure is recorded as a percentage(0-100%) and the normal range is 50-85%.
  LV Fractional Shortening is the percent change in a patient's LV internal dimensions between systole (when the ventricles contract and expel blood) and diastole (when the ventricles expand and receive blood). The measure is recorded as a percentage(0-100%) and the normal range is 30-45%.
Time Frame: Baseline, 12, and 24 month visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of LV unit
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
percentage of LV unit
  LV Fractional Shortening (%) at Baseline | 19.5 (9.2) | 18.8 (8.5)
  LV Fractional Shortening (%) at 12 Months | 21.6 (8.4) | 20.1 (8.0)
  LV Fractional Shortening (%) at 24 Months | 21.3 (9.1) | 20.6 (8.6)
  LV Ejection Fraction (%) at Baseline | 35.3 (11.9) | 35.5 (11.6)
  LV Ejection Fraction (%) at 12 Months | 38.8 (11.9) | 37.3 (11.8)
  LV Ejection Fraction (%) at 24 Months | 37.6 (12.5) | 36.7 (12.0)
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; A linear mixed model was fit for each of the following: LV Ejection Fraction and LV Fractional Shortening; the purpose was to test whether patients with MVP and no pacing indication over time had a different average value for that measure than patients with VVI and no pacing indication. Two-sided tests were used. Data were also collected from the 36 month visits but were excluded due to the trial being stopped early and only a subset of patients having data for those visits; Test type: Superiority or Other; p > 0.10, Mixed Models Analysis — The a priori threshold for significance for Arm was 0.05, with no adjustment for multiple analyses; Models were fit with time and arm as covariates

6. Secondary Outcome: Left Ventricular (LV) and Left Atrial (LA) Volumes
Description: Echocardiogram measures for each endpoint were obtained at multiple time points.
Time Frame: Baseline, 12, and 24 month visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
milliliters (mL)
  LV End Systolic Volume (LVESV) at Baseline | 127.6 (65.5) | 121.2 (54.4)
  LVESV at 12 Months | 108.9 (59.7) | 105.8 (53.4)
  LVESV at 24 Months | 116.5 (62.6) | 108.7 (52.8)
  LV End Diastolic Volume (LVEDV) at Baseline | 189.8 (72.7) | 182.5 (60.6)
  LVEDV at 12 Months | 170.6 (68.6) | 163.2 (58.7)
  LVEDV at 24 Months | 179.0 (71.8) | 165.8 (57.8)
  Left Atrial (LA) Volume at Baseline | 75.4 (26.1) | 74.5 (26.5)
  LA Volume at 12 Months | 74.5 (28.3) | 73.6 (27.9)
  LA Volume at 24 Months | 82.3 (32.0) | 77.4 (27.7)
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; A linear mixed model was fit to test whether patients with MVP and no pacing indication had a different values for left ventricular end diastolic volume ("LVEDV") over time than similar patients with VVI 40. A two-sided test was used. Data were collected from the 36 month visits but were excluded due to the trial being stopped early and only a subset of patients having data for those visits; Test type: Superiority or Other; p = 0.0424, Mixed Models Analysis — The a priori threshold for statistical significance for Arm was 0.05, with no correction for multiple comparisons; The model was fit with time and arm as covariates
Statistical Analysis 2: Comparison: VVI 40 vs MVP Pacing; Similar models were fit for left ventricle ("LV") End Systolic Volume and Left Atrial Volume; Test type: Superiority or Other; p > 0.10, Mixed Models Analysis — In each case the a priori threshold for significance for Arm was 0.05; Models were fit with time and arm as covariates

7. Secondary Outcome: Left Ventricular (LV) Sphericity Index
Description: Echocardiogram measures for each endpoint were obtained at multiple time points.
  LV Sphericity Index is a ratio of LV long axis dimension to the LV short axis dimension. Healthy hearts have an elliptical LV cross-sectional shape. A value of 1 denotes a circular or more globular shape, while larger values denote healthier hearts with more elliptical cross sections. Literature has shown that when the ratio used is short axis/long axis, normal hearts have a median LV sphericity index of 0.56, with a range of (0.51-0.60). This translates to median=1.79,range=(1.67,1.96) for long/short axis.
Time Frame: Baseline, 12, and 24 month visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
Ratio
  Left Ventricular (LV) Sphericity Index at Baseline | 1.5 (0.2) | 1.5 (0.2)
  LV Sphericity Index at 12 Months | 1.5 (0.2) | 1.5 (0.2)
  LV Sphericity Index at 24 Months | 1.6 (0.2) | 1.5 (0.2)
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; A linear mixed model was fit to test whether patients with MVP and no pacing indication had a different values of Left Ventricular Sphericity Index over time than similar patients with VVI 40. A two-sided test was used. Data were collected from the 36 month visits but were excluded due to the trial being stopped early and only a subset of patients having data for those visits; Test type: Superiority or Other; p = 0.0418, Mixed Models Analysis — The a priori threshold for significance for Arm was 0.05, with no adjustment for multiple analyses; The model fit with time and arm as covariates

8. Secondary Outcome: Hemodynamic Velocity Measures
Description: Echocardiogram measures for each endpoint were obtained at multiple time points.
Time Frame: Baseline, 12, and 24 month visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
meters per second (m/s)
  Tricuspid Regurgitation (TR) Velocity at Baseline | 2.7 (0.4) | 2.7 (0.5)
  TR Velocity at 12 Months | 2.7 (0.4) | 2.7 (0.4)
  TR Velocity at 24 Months | 2.7 (0.4) | 2.6 (0.5)
  Mitral Inflow - peak E at Baseline | 0.8 (0.2) | 0.8 (0.3)
  Mitral Inflow - peak E at 12 Months | 0.7 (0.3) | 0.7 (0.3)
  Mitral Inflow - peak E at 24 Months | 0.7 (0.3) | 0.7 (0.3)
  Mitral Inflow - peak A at Baseline | 0.7 (0.3) | 0.7 (0.3)
  Mitral Inflow - peak A at 12 Months | 0.7 (0.2) | 0.8 (0.2)
  Mitral Inflow - peak A at 24 Months | 0.7 (0.2) | 0.8 (0.2)
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; A linear mixed model was fit for each of the following: TR Velocity, Mitral Inflow-peak E and Mitral Inflow-peak A; the purpose was to test whether patients with MVP and no pacing indication over time had a different average value for that measure than patients with VVI and no pacing indication. Two-sided tests were used. Data were collected from the 36 month visits but were excluded due to the trial being stopped early and only a subset of patients having data for those visits; Test type: Superiority or Other; p > 0.10, Mixed Models Analysis — The a priori threshold for statistical significance for Arm was 0.05, with no correction for multiple comparisons; Models were fit with time and arm as covariates

9. Secondary Outcome: Hemodynamic Deceleration Time
Description: Echocardiogram measures for each endpoint were obtained at multiple time points.
Time Frame: Baseline, 12, and 24 month visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
milliseconds (ms)
  Mitral Inflow - Deceleration Time at Baseline | 194.6 (50.6) | 192.3 (50.6)
  Mitral Inflow - Deceleration Time at 12 Months | 206.8 (54.7) | 208.7 (61.0)
  Mitral Inflow - Deceleration Time at 24 Months | 208.0 (54.6) | 210.7 (56.9)
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; A linear mixed model was fit for Mitral Inflow - Deceleration time; the purpose was to test whether patients with MVP and no pacing indication over time had a different average value for that measure than patients with VVI and no pacing indication. A two-sided test was used. Data were collected from the 36 month visits but were excluded due to the trial being stopped early and only a subset of patients having data for those visits; Test type: Superiority or Other; p = 0.9490, Mixed Models Analysis — The a priori threshold for significance for Arm was 0.05, with no adjustment for multiple analyses; Model fit with time and arm as covariates

10. Secondary Outcome: Left Atrial (LA) and Mitral Regurgitation (MR) Areas
Description: Echocardiogram measures for each endpoint were obtained at multiple time points.
Time Frame: Baseline, 12, and 24 month visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters squared (cm2)
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
centimeters squared (cm2)
  Left Atrial (LA) Area at Baseline | 22.7 (5.8) | 22.5 (5.9)
  LA Area at 12 Months | 22.0 (5.5) | 21.9 (6.4)
  LA Area at 24 Months | 22.0 (6.0) | 21.9 (6.3)
  Mitral Regurgitation (MR) Area at Baseline | 4.8 (4.3) | 5.1 (4.7)
  MR Area at 12 Months | 4.8 (4.9) | 4.5 (4.3)
  MR Area at 24 Months | 5.0 (4.5) | 4.7 (4.0)
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; A linear mixed model was fit for each of the following: Left Atrial Area and Mitral Regurgitation Area; the purpose was to test whether patients with MVP and no pacing indication over time had a different average value for that measure than patients with VVI and no pacing indication. Two-sided tests were used. Data were collected from the 36 month visits but were excluded due to the trial being stopped early and only a subset of patients having data for those visits; Test type: Superiority or Other; p > 0.10, Mixed Models Analysis — The a priori threshold for significance for Arm was 0.05, with no adjustment for multiple analyses; Models fit with time and arm as covariates

11. Secondary Outcome: Composite Mitral Regurgitation (MR) Severity Score
Description: Echocardiogram measures for this endpoint were obtained at multiple time points. Composite MR Severity was measured on a scale of "None to Trivial" to "Grade IV", with Grade IV being the worst possible score and "None to Trivial" being the best possible score.
Time Frame: Baseline, 12, and 24 month visits
Measure: Number; unit: participants
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
participants
  Baseline MR Score of None to Trivial | 236 | 232
  Baseline MR Score: Grade I | 160 | 148
  Baseline MR Score: Grade II | 48 | 63
  Baseline MR Score: Grade III | 18 | 14
  Baseline MR Score: Grade IV | 10 | 14
  Baseline MR Score: Indeterminate | 9 | 22
  12 Month MR Score: None to Trivial | 198 | 201
  12 Month MR Score: Grade I | 133 | 119
  12 Month MR Score: Grade II | 46 | 42
  12 Month MR Score: Grade III | 17 | 13
  12 Month MR Score: Grade IV | 6 | 4
  12 Month Score: Indeterminate | 8 | 14
  24 Month MR Score: None to Trivial | 174 | 164
  24 Month MR Score: Grade I | 130 | 118
  24 Month MR Score: Grade II | 30 | 27
  24 Month MR Score: Grade III | 8 | 11
  24 Month MR Score: Grade IV | 9 | 6
  24 Month Score: Indeterminate | 6 | 9
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; A General Estimating Equation ("GEE") Cumulative Logits model was fit with Arm, Time, and their interaction as covariates in the model to test the hypothesis that patients with no pacing indication and MVP programming have different Mitral Regurgation over time than similar patients with VVI 40 programming. A two-sided test was used. Data were collected from the 36 month visits but were excluded due to the trial being stopped early and only a subset of patients having data for those visits; Test type: Superiority or Other; p = 0.8403, Cumulative Logits Model — The a priori threshold for significance for Arm was 0.05; Because Composite Mitral Regurgitation Score was measured on the ordinal scale, a GEE cumulative logits model was fit

12. Secondary Outcome: Occurrence of Ventricular Tachycardia ("VT") and Ventricular Fibrillation ("VF") Episodes
Description: Annualized Rates of Days of True VT/VF and Inappropriately detected non-VT/VF
Time Frame: Enrollment to last collection of data from the implanted ICD (up to 45 months post-randomization)
Population: as for outcome 1
Measure: Number; unit: Annualized Episodes per Patient Month
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
Annualized Episodes per Patient Month
  True VT/VF | 0.170 | 0.155
  Inappropriately detected non-VT/VF | 0.038 | 0.055
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; The pre-specified analysis called for a comparison of the hazard rates of true VT/VF between the two arms by way of a one-sided 95% confidence interval on the hazard ratio (values less than one favor MVP) after fitting a model. The unit of time was days, not episodes, so the analysis did not account for multiple episodes on the same day. If the upper bound was less than 1, the null hypothesis of equal hazard rates would be rejected; Test type: Superiority or Other; Andersen-Gill model; This model was fit to account for multiple events (i.e. days in which true VT/VF occurred) within subject; Hazard Ratio (HR) = 0.949, 95% CI [0.949 to 1.209] — Because of the possible correlation within subject of days with episodes, a subsequent analysis was done using a bootstrap confidence interval for the annualized rate of episodes per patient month
Statistical Analysis 2: Comparison: VVI 40 vs MVP Pacing; A 95% one-sided bootstrap confidence interval was generated for the MVP - VVI 40 difference in annualized rates of true VT/VF per patient month. If the interval upper bound was less than 0, the null hypothesis of equal rates would be rejected; Test type: Superiority or Other; Bootstrap Confidence Interval; Difference in Annualized Rates = -0.015, 95% CI [-0.015 to 0.033]
Statistical Analysis 3: Comparison: VVI 40 vs MVP Pacing; The pre-specified analysis called for a comparison of the hazard rates of inappropriately detected non-VT/VF between the two arms by way of a one-sided 95% confidence interval on the hazard ratio (MVP in numerator) after fitting a model. The unit of time was days, not episodes, so the analysis did not account for multiple episodes on the same day. If the upper bound was less than 1, the null hypothesis of equal hazard rates would be rejected; Test type: Superiority or Other; Andersen-Gill model; This model was fit to account for multiple events (i.e. days in which non-VT/VF detected by device as VT/VF) within subject; Hazard Ratio (HR) = 1.310, 95% CI [1.310 to 1.858] — Because of the possible correlation within a subject for days with episodes, a subsequent analysis was done using a bootstrap confidence interval for the annualized rate of episodes per patient month
Statistical Analysis 4: Comparison: VVI 40 vs MVP Pacing; A 95% one-sided bootstrap confidence interval was generated for the MVP - VVI 40 difference in annualized rates of inappropriately detected non-VT/VF per patient month. If the interval upper bound was less than 0, the null hypothesis of equal rates would be rejected; Test type: Superiority or Other; Bootstrap Confidence Interval; Difference in Annualized Rates = 0.017, 95% CI [0.017 to 0.036]

13. Secondary Outcome: Occurrence of Clinically Important or Persistent Atrial Tachycardia or Atrial Fibrillation (AT/AF) in Subjects With no Prior AF History
Description: Persistent AF was defined as any of the following:
  1. 2 consecutive visits in which the patient presents with AF
  2. 7 consecutive days of at least 22 hours per day of AT/AF
  3. A cardioversion prior to 7 consecutive days of at least 22 hours per day of AT/AF
  Clinically Important AF was defined as more than 20 hours of AT/AF in a single day
Time Frame: Enrollment to last collection of data from the implanted ICD (up to 45 months post-randomization)
Population: 1 of 1031 randomized subjects had a history of at least 6 months of chronic AF, which was an exclusion criterion. Of the remaining 1030 randomized subjects that met all inclusion criteria, only those with no history of AF were included in the analysis (445 in the VVI 40 arm and 444 in the MVP arm). An intention to treat analysis was performed.
Measure: Number; unit: participants
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
participants | 445 | 444
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; This analysis compared the hazard rates for clinically important AF (defined as a calendar day with >20 hour of AT/AF as measured by the device). The null hypothesis was that this hazard rate for patients with MVP was equal to or greater than that of patients with VVI 40. The pre-specified model had Arm as a covariate, and accounted for time to first event and time between successive events per subject; Test type: Superiority or Other; p = 0.7166, Andersen-Gill model — The threshold for significance was the one-sided upper confidence bound being less than 1; Hazard Ratio (HR) = 1.22, 95% CI [1.22 to 3.0]
Statistical Analysis 2: Comparison: VVI 40 vs MVP Pacing; This analysis compared the percentage of days with >20 hours of AT/AF as measured by the device(definition of clinically important AF) between arms. The null hypothesis was that this percentage of days for patients with MVP was equal or greater to that of patients with VVI 40; Test type: Superiority or Other; Bootstrap Confidence Interval — The threshold for significance was defined as the upper one-sided confidence bound being less than 0; Mean Difference (Net) = 0.15, 95% CI 2-sided [-100 to 0.8]
Statistical Analysis 3: Comparison: VVI 40 vs MVP Pacing; This analysis tested the null hypothesis that the hazard rate for development of persistent AF(defined as 2 consecutive visits presenting with AT/AF, 7 consecutive days of 22 or more hours per day of AT/AF, or < 7 such days due to a cardioversion) in patients with MVP and no pacing indication was equal to or greater than that of similar patients with VVI 40; Test type: Superiority or Other; p = 0.325, Log Rank — The a priori threshold for statistical significance was 0.05; A one-sided test was used
Statistical Analysis 4: Comparison: VVI 40 vs MVP Pacing; This analysis tested the hypothesis that the average AT/AF burden (hours per day of AT/AF) through 6 months post-implant in patients with no Class I pacing indication and MVP is equal to or greater than that of similar patients with VVI 40. Only subjects with complete AT/AF data for this time interval were included in the analysis; Test type: Superiority or Other; Bootstrap Confidence Interval — The a priori threshold for significance was defined as the one-sided upper 95% confidence bound for the MVP - VVI 40 difference in average AT/AF through 6 months being less than 0; Mean Difference (Final Values) = 0, 95% CI [0 to 0.145]
Statistical Analysis 5: Comparison: VVI 40 vs MVP Pacing; This analysis tested the hypothesis that the average AT/AF burden (hours per day of AT/AF) from 6 to 12 months post-implant in patients with no Class I pacing indication and MVP is equal to or greater than that of similar patients with VVI 40. Only subjects with complete AT/AF data for this time interval were included in the analysis; Test type: Superiority or Other; Bootstrap Confidence Interval — The a priori threshold for significance was defined as the one-sided upper 95% confidence bound for the MVP - VVI 40 difference in average AT/AF burden from 6 to 12 months being less than 0; Mean Difference (Final Values) = 0, 95% CI [0 to 0.227]
Statistical Analysis 6: Comparison: VVI 40 vs MVP Pacing; This analysis tested the hypothesis that the average AT/AF burden (hours per day of AT/AF) from 12 to 24 months post-implant in patients with no Class I pacing indication and MVP is equal to or greater than that of similar patients with VVI 40. Only subjects with complete AT/AF data for this time interval were included in the analysis; Test type: Superiority or Other; Bootstrap Confidence Interval — The a priori threshold for significance was defined as the one-sided upper 95% confidence bound for the MVP - VVI 40 difference in average AT/AF burden from 12 to 24 months being less than 0; Mean Difference (Final Values) = 0, 95% CI [0 to 0.261]
Statistical Analysis 7: Comparison: VVI 40 vs MVP Pacing; This analysis tested the hypothesis that the average AT/AF burden (hours per day of AT/AF) from 24 to 36 months post-implant in patients with no Class I pacing indication and MVP is equal to or greater than that of similar patients with VVI 40. Only subjects with complete AT/AF data for this time interval were included in the analysis; Test type: Superiority or Other; Bootstrap Confidence Interval — The a priori threshold for significance was defined as the one-sided upper 95% confidence bound for the MVP - VVI 40 difference in average AT/AF burden from 24 to 36 months being less than 0; Mean Difference (Final Values) = -0.1, 95% CI [-0.1 to 0.110]

14. Secondary Outcome: Development of a Pacing Indication During the Study
Description: Physician identification of a Class I Pacing Indication. A Class I Pacing Indication implies that the benefit of pacing the heart far exceeds the risk, and that the procedure to implant the pacing device should be performed. For this indication there is general agreement that pacing the heart is beneficial, useful, and effective.
Time Frame: Enrollment to last visit (up to 45 months post-randomization)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
participants | 38 | 19
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; Physicians recorded at each scheduled and unscheduled follow-up whether the subject had developed a Class I indication since their last visit. The time from randomization to Class I indication development or last visit if censored was determined for each subject. The null hypothesis was that the hazard rate for time to development of a Class I pacing indication among patients with MVP programming was equal to or greater than that of patients with VVI 40 programming; Test type: Superiority or Other; p = 0.0053, Log Rank — The a priori threshold for statistical significance was 0.05. The threshold was met, and the null hypothesis rejected

15. Secondary Outcome: Medication Usage Affecting Heart Rate and Atrioventricular ("AV") Conduction
Description: Whether a subject is on each of a pre-specified set of drugs or classes of drugs.
Time Frame: Enrollment, 6 Months, 12 Months, 24 Months, 30 Months, 36 Months
Population: as for outcome 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
Percentage of Subjects
  Baseline Amiodarone | 12.7 | 11.4
  6 Month Amiodarone | 12.2 | 12.4
  12 Month Amiodarone | 12.5 | 13.1
  24 Month Amiodarone | 12.7 | 14.8
  30 Month Amiodarone | 13.5 | 12.1
  36 Month Amiodarone | 8.0 | 12.3
  Baseline Sotalol | 1.0 | 0.8
  6 Month Sotalol | 1.4 | 1.6
  12 Month Sotalol | 2.0 | 1.0
  24 Month Sotalol | 2.7 | 1.4
  30 Month Sotalol | 3.6 | 3.0
  36 Month Sotalol | 5.3 | 1.4
  Baseline Beta Blockers | 88.7 | 88.4
  6 Month Beta Blockers | 91.1 | 90.6
  12 Month Beta Blockers | 92.3 | 90.3
  24 Month Beta Blockers | 92.6 | 90.2
  30 Month Beta Blockers | 91.0 | 92.9
  36 Month Beta Blockers | 89.3 | 87.7
  Baseline Amlodipine | 5.5 | 6.6
  6 Month Amlodipine | 4.9 | 7.3
  12 Month Amlodipine | 5.7 | 7.4
  24 Month Amlodipine | 6.6 | 8.4
  30 Month Amlodipine | 7.2 | 9.1
  36 Month Amlodipine | 6.7 | 13.7
  Baseline Diltiazem | 1.8 | 0.6
  6 Month Diltiazem | 1.9 | 0.7
  12 Month Diltiazem | 1.8 | 0.7
  24 Month Diltiazem | 1.9 | 0.6
  30 Month Diltiazem | 1.8 | 0
  36 Month Diltiazem | 2.7 | 1.4
  Baseline Verapamil | 0.8 | 0.4
  6 Month Verapamil | 1.2 | 0.5
  12 Month Verapamil | 0.7 | 0.5
  24 Month Verapamil | 1.6 | 0.3
  30 Month Verapamil | 0 | 0
  36 Month Verapamil | 4.0 | 0
  Baseline ACE-Inhibitors | 66.7 | 68.9
  6 Month ACE-Inhibitors | 64.9 | 70.7
  12 Month ACE-Inhibitors | 67.6 | 70.8
  24 Month ACE-Inhibitors | 67.6 | 70.7
  30 Month ACE-Inhibitors | 73.0 | 74.7
  36 Month ACE-Inhibitors | 70.7 | 64.4
  Baseline ARBs | 18.1 | 15.4
  6 Month ARBs | 20.7 | 16.4
  12 Month ARBs | 20.9 | 17.3
  24 Month ARBs | 21.8 | 17.9
  30 Month ARBs | 19.8 | 17.2
  36 Month ARBs | 20.0 | 26.0
  Baseline Aldosterone Receptor Antagonists | 17.9 | 19.1
  6 Month Aldosterone Receptor Antagonists | 17.6 | 21.3
  12 Month Aldosterone Receptor Antagonists | 17.9 | 21.4
  24 Month Aldosterone Receptor Antagonists | 16.4 | 21.5
  30 Month Aldosterone Receptor Antagonists | 17.1 | 24.2
  36 Month Aldosterone Receptor Antagonists | 13.3 | 17.8
  Baseline Spironolactone | 13.8 | 13.3
  6 Month Spironolactone | 13.2 | 15.2
  12 Month Spironolactone | 13.4 | 14.3
  24 Month Spironolactone | 13.3 | 15.1
  30 Month Spironolactone | 16.2 | 17.2
  36 Month Spironolactone | 10.7 | 12.3
  Baseline Diuretics | 54.2 | 53.9
  6 Month Diuretics | 58.6 | 56.4
  12 Month Diuretics | 58.0 | 57.2
  24 Month Diuretics | 58.6 | 58.1
  30 Month Diuretics | 56.8 | 56.6
  36 Month Diuretics | 56.0 | 60.3
  Baseline Digoxin | 21.6 | 18.7
  6 Month Digoxin | 21.6 | 17.8
  12 Month Digoxin | 21.5 | 18.5
  24 Month Digoxin | 20.4 | 17.9
  30 Month Digoxin | 22.5 | 19.2
  36 Month Digoxin | 17.3 | 8.2

16. Secondary Outcome: Percent Ventricular Pacing
Description: The percentage of a patients' ventricular beats that were paced by the device.
Time Frame: Enrollment, 6, 12, 24 and 36 month visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent pacing
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
Percent pacing
  Baseline to 6 Months | 0.7 (3.7) | 0.8 (3.4)
  Baseline to 12 Months | 1.1 (5.5) | 1.0 (4.0)
  Baseline to 24 Months | 1.8 (8.0) | 1.6 (6.4)
  Baseline to 36 Months | 3.4 (13.8) | 1.5 (6.9)
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; All subjects from the analysis cohort with available data for the time period of interest were included in the corresponding analysis. The null hypothesis was that the average percent ventricular pacing through 6 months post-implant for patients with MVP programming and was greater than or equal to that of patients with VVI 40 programming; Test type: Superiority or Other; p = 0.9791, Wilcoxon (Mann-Whitney) — The one-sided Wilcoxon Rank Sum test yielded a p-value greater than 0.05, which was the a priori threshold for significance
Statistical Analysis 2: Comparison: VVI 40 vs MVP Pacing; All subjects from the analysis cohort with available data for the time period of interest were included in the corresponding analysis. The null hypothesis was that the average percent ventricular pacing through 12 months post-implant for patients with MVP programming was greater than or equal to that of patients with VVI 40 programming; Test type: Superiority or Other; p = 0.8984, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 16, analysis 1]; Alternative hypothesis:patients with MVP & no pacing indication have less mean ventricular pacing through 12 months than similar patients with VVI 40
Statistical Analysis 3: Comparison: VVI 40 vs MVP Pacing; All subjects from the analysis cohort with available data for the time period of interest were included in the corresponding analysis. The null hypothesis was that the average percent ventricular pacing through 24 months post-implant for patients with MVP programming and no pacing indication was greater than or equal to that of patients with VVI 40 programming and no pacing indication; Test type: Superiority or Other; p = 0.7144, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 16, analysis 1]; Alternative hypothesis:patients with MVP & no pacing indication have less mean ventricular pacing through 24 months than similar patients with VVI 40
Statistical Analysis 4: Comparison: VVI 40 vs MVP Pacing; All subjects from the analysis cohort with available data for the time period of interest were included in the corresponding analysis. The null hypothesis was that the average percent ventricular pacing through 36 months post-implant for patients with MVP programming and no pacing indication was greater than or equal to that of patients with VVI 40 programming and no pacing indication; Test type: Superiority or Other; p = 0.5165, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 16, analysis 1]; Alternative hypothesis:patients with MVP & no pacing indication have less mean ventricular pacing through 36 months than similar patients with VVI 40

17. Secondary Outcome: Quality of Life ("QOL") Score
Description: Minnesota Living with Heart Failure Questionnaire ("MLWHFQ") and Kansas City Cardiomyopathy Questionnaire ("KCCQ") Quality of Life("QOL") Scores. For KCCQ, positive values mean improved QOL compared to baseline. For MLWHFQ, negative values mean improved QOL compared to baseline.
  Scales: KCCQ 0-100 (0=worst, 100 best); MLWHFQ 0-105 (105=worst, 0=best)
Time Frame: Baseline, 12, 24, and 36 month visits
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
Units on a scale
  KCCQ Physical Limitation(12 Mo. -Baseline Change) | 0.3 (25.8) | 4.1 (28.5)
  KCCQ Physical Limitation(24 Mo. -Baseline Change) | -2.2 (28.5) | -0.1 (31.4)
  KCCQ Physical Limitation(36 Mo. -Baseline Change) | -11.0 (32.5) | -11.0 (30.8)
  KCCQ Symptom Stability(12 Mo. -Baseline Change) | 1.8 (28.5) | 3.1 (27.1)
  KCCQ Symptom Stability(24 Mo. -Baseline Change) | -1.5 (28.5) | -0.6 (30.7)
  KCCQ Symptom Stability(36 Mo. -Baseline Change) | -10.8 (29.0) | -10.5 (33.6)
  KCCQ Symptom Frequency(12 Mo. -Baseline Change) | 4.7 (27.8) | 5.1 (27.4)
  KCCQ Symptom Frequency(24 Mo. -Baseline Change) | 2.2 (31.9) | 1.7 (31.8)
  KCCQ Symptom Frequency(36 Mo. -Baseline Change) | -7.1 (37.4) | -10.1 (33.1)
  KCCQ Symptom Burden(12 Mo. -Baseline Change) | 4.8 (27.7) | 5.9 (28.6)
  KCCQ Symptom Burden(24 Mo. -Baseline Change) | 2.4 (32.3) | 3.2 (33.0)
  KCCQ Symptom Burden(36 Mo. -Baseline Change) | -7.3 (38.2) | -8.6 (34.3)
  KCCQ Total Symptoms(12 Mo. -Baseline Change) | 4.7 (26.7) | 5.5 (26.9)
  KCCQ Total Symptoms(24 Mo. -Baseline Change) | 2.3 (31.2) | 2.4 (31.4)
  KCCQ Total Symptoms(36 Mo. -Baseline Change) | -7.2 (36.9) | -9.3 (33)
  KCCQ Self-Efficacy(12 Mo. -Baseline Change) | 1.9 (28.9) | 4.9 (30.5)
  KCCQ Self-Efficacy(24 Mo. -Baseline Change) | -0.9 (34.1) | -0.2 (35.9)
  KCCQ Self-Efficacy(36 Mo. -Baseline Change) | -12.6 (43.2) | -12.5 (43.5)
  KCCQ Quality of Life(12 Mo. -Baseline Change) | 12.9 (31.8) | 16.6 (32.1)
  KCCQ Quality of Life(24 Mo. -Baseline Change) | 11.3 (35.7) | 14.6 (35.5)
  KCCQ Quality of Life(36 Mo. -Baseline Change) | 0.7 (39.4) | 0.9 (33.1)
  KCCQ Social Limitation(12 Mo.-Baseline Change) | 5.6 (31.7) | 8.1 (33.5)
  KCCQ Social Limitation(24 Mo.-Baseline Change) | 3.4 (35.9) | 6.1 (36.4)
  KCCQ Social Limitation(36 Mo.-Baseline Change) | -6.4 (40.7) | -2.3 (32.2)
  KCCQ Overall Summary(12 Mo.-Baseline Change) | 6.1 (25.1) | 8.7 (26.7)
  KCCQ Overall Summary(24 Mo.-Baseline Change) | 3.7 (29.4) | 5.7 (30.2)
  KCCQ Overall Summary(36 Mo.-Baseline Change) | -5.1 (34.7) | -5.4 (28.7)
  KCCQ Clinical Summary(12 Mo.-Baseline Change) | 2.8 (24.1) | 4.9 (25.9)
  KCCQ Clinical Summary(24 Mo.-Baseline Change) | 0.2 (28.1) | 1.2 (29.3)
  KCCQ Clinical Summary(36 Mo.-Baseline Change) | -8.4 (33.8) | -9.7 (29.6)
  MLWHFQ (12 Month - Baseline Change) | -5.8 (24.6) | -7.9 (28.5)
  MLWHFQ (24 Month - Baseline Change) | -2 (30.6) | -4 (31.7)
  MLWHFQ (36 Month - Baseline Change) | 8.4 (37) | 5.9 (32.1)
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; For the KCCQ Physical Limitation Score, the change from baseline to 12 months was compared between the two arms, using a two-sided test. If a subject died prior to the time point, a score of 0 was imputed for their 12 month score; Test type: Superiority or Other; p = 0.0073, Wilcoxon (Mann-Whitney) — The p-value is not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: VVI 40 vs MVP Pacing; For the KCCQ Symptom Stability Score, the change from baseline to 12 months was compared between the two arms, using a two-sided test. If a subject died prior to the time point, a score of 0 was imputed for their 12 month score; Test type: Superiority or Other; p = 0.2493, Wilcoxon (Mann-Whitney) — No adjustment was made for multiple comparisons, and the a priori threshold for statistical significance was 0.05
Statistical Analysis 3: Comparison: VVI 40 vs MVP Pacing; For the KCCQ Symptom Frequency Score, the change from baseline to 12 months was compared between the two arms, using a two-sided test. If a subject died prior to the time point, a score of 0 was imputed for their 12 month score; Test type: Superiority or Other; p = 0.7728, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, and no adjustment was made for multiple comparisons
Statistical Analysis 4: Comparison: VVI 40 vs MVP Pacing; For the KCCQ Symptom Burden Score, the change from baseline to 12 months was compared between the two arms, using a two-sided test. If a subject died prior to the time point, a score of 0 was imputed for their 12 month score; Test type: Superiority or Other; p = 0.3082, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, and no adjustment was made for multiple comparisons
Statistical Analysis 5: Comparison: VVI 40 vs MVP Pacing; For the KCCQ Total Symptom Score, the change from baseline to 12 months was compared between the two arms, using a two-sided test. If a subject died prior to the time point, a score of 0 was imputed for their 12 month score; Test type: Superiority or Other; p = 0.5422, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, and no adjustment was made for multiple comparisons
Statistical Analysis 6: Comparison: VVI 40 vs MVP Pacing; For the KCCQ Self-Efficacy Score, the change from baseline to 12 months was compared between the two arms, using a two-sided test. If a subject died prior to the time point, a score of 0 was imputed for their 12 month score; Test type: Superiority or Other; p = 0.0851, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, and no adjustment was made for multiple comparisons
Statistical Analysis 7: Comparison: VVI 40 vs MVP Pacing; For the KCCQ Quality of Life Score, the change from baseline to 12 months was compared between the two arms, using a two-sided test. If a subject died prior to the time point, a score of 0 was imputed for their 12 month score; Test type: Superiority or Other; p = 0.0502, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, and no adjustment was made for multiple comparisons
Statistical Analysis 8: Comparison: VVI 40 vs MVP Pacing; For the KCCQ Social Limitation Score, the change from baseline to 12 months was compared between the two arms, using a two-sided test. If a subject died prior to the time point, a score of 0 was imputed for their 12 month score; Test type: Superiority or Other; p = 0.0463, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, and no adjustment was made for multiple comparisons
Statistical Analysis 9: Comparison: VVI 40 vs MVP Pacing; For the KCCQ Overall Summary Score, the change from baseline to 12 months was compared between the two arms, using a two-sided test. If a subject died prior to the time point, a score of 0 was imputed for their 12 month score; Test type: Superiority or Other; p = 0.0227, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, and no adjustment was made for multiple comparisons
Statistical Analysis 10: Comparison: VVI 40 vs MVP Pacing; For the KCCQ Overall Clinical Summary Score, the change from baseline to 12 months was compared between the two arms, using a two-sided test. If a subject died prior to the time point, a score of 0 was imputed for their 12 month score; Test type: Superiority or Other; p = 0.0582, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, and no adjustment was made for multiple comparisons
Statistical Analysis 11: Comparison: VVI 40 vs MVP Pacing; The 10 KCCQ analyses were repeated comparing changes from baseline to 24 months between arms. Again if a subject died prior to their 24 month visit, a value of 0 was imputed for their 24 month score; Test type: Superiority or Other; p > 0.15, Wilcoxon (Mann-Whitney) — Tests for all ten KCCQ subscores yielded p-values greater than 0.15 (the a priori threshold for statistical significance was 0.05)
Statistical Analysis 12: Comparison: VVI 40 vs MVP Pacing; The 10 KCCQ analyses were repeated comparing changes from baseline to 36 months between arms. Again if a subject died prior to their 36 month visit, a value of 0 was imputed for their 36 month score; Test type: Superiority or Other; p > 0.15, Wilcoxon (Mann-Whitney) — Tests for all 10 KCCQ subscores yielded p-values greater than 0.15 (the a priori threshold for statistical significance was 0.05); Because the trial was stopped early, only 178 subjects were included in these analyses
Statistical Analysis 13: Comparison: VVI 40 vs MVP Pacing; The change in Minnesota Living with Heart Failure Questionnaire score from baseline to 12 months was compared using a two-sided test. If a subject died before their 12 month visit, a value of 105 (worst possible MLWHF score) was imputed for their 12 month score; Test type: Superiority or Other; p = 0.1399, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, and no adjustment was made for multiple comparisons
Statistical Analysis 14: Comparison: VVI 40 vs MVP Pacing; The change in Minnesota Living with Heart Failure Questionnaire score from baseline to 24 months was compared using a two-sided test. If a subject died before their 24 month visit, a value of 105 (worst possible MLWHF score) was imputed for their 24 month score; Test type: Superiority or Other; p = 0.3573, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, and no adjustment was made for multiple comparisons
Statistical Analysis 15: Comparison: VVI 40 vs MVP Pacing; The change in Minnesota Living with Heart Failure Questionnaire score from baseline to 36 months was compared using a two-sided test. If a subject died before their 36 month visit, a value of 105 (worst possible MLWHF score) was imputed for their 36 month score; Test type: Superiority or Other; p = 0.5183, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was 0.05, with no adjustment made for multiple comparisons; Because the trial was stopped early, only 178 subjects were included in this analysis

18. Secondary Outcome: All Cause Mortality
Description: Death from any cause
Time Frame: Enrollment to last visit (up to 45 months post-randomization) or death
Population: as for outcome 1
Measure: Number; unit: participants who died
Arm/Group | VVI 40 | MVP Pacing
Number analyzed (Participants) | 512 | 518
participants who died | 46 | 57
Statistical Analysis 1: Comparison: VVI 40 vs MVP Pacing; The time from randomization to all cause mortality or last follow-up visit was determined for each subject. The null hypothesis was that the mortality hazard rate for patients with MVP programming was greater than that of patients with VVI40 programming; Test type: Non-Inferiority or Equivalence — A non-inferiority analysis was performed, with the hazard ratio as the parameter of interest and the non-inferiority threshold of 1.44. The one-sided upper confidence bound for the hazard ratio had to be less than 1.44 for the null hypothesis to be rejected. The threshold of 1.44 was derived by using a noninferiority threshold of a 5 percentage point difference in 24 month survival rates; Hazard Ratio (HR) = 1.26, 95% CI [1.26 to 1.75] — This was a non-inferiority analysis, and so a one-sided 95% confidence interval was performed comparing the MVP arm to the VVI 40 arm

19. Secondary Outcome: ICD-indicated Patients With Class I Pacemaker Indication.
Description: Number of subjects screened prior to enrollment that had Class I pacing indication at time of implant
Time Frame: Period of time prior to patient consent when considering patient for Implant/Enrollment
Population: Centers kept a screening log, recording for each patient considered for new ICD implant and possible trial enrollment whether the patient had a Class I pacing indication at time of implant. The analysis consisted of descriptive statistics (counts of the 2051 screened patients).
Measure: Number; unit: participants
Groups:
- All Screened Patients: All Patients Screened for Possible Enrollment
Arm/Group | All Screened Patients
Number analyzed (Participants) | 2051
participants
  Class I Pacing Indication at Implant | 220 (0.68)
  No Class I Pacing Indication at Implant | 1818 (0.70)
  Class I Pacing Indication Status Not Recorded | 13 (2.20)

ADVERSE EVENTS:
Time Frame: From enrollment to study exit or closure (up to 45 months post-randomization)
Description: Adverse Events defined as any undesirable clinical occurrence in a subject. Data collection limited to cardiovascular, pulmonary or renal system (including system and procedure-related events) or events in which the subject presented with symptoms compatible with fluid retention and/or decreased exercise tolerance.
Arm/Group | VVI 40 Pacing | MVP Pacing
Serious Adverse Events (participants affected / at risk) | 128/513 | 121/518
Other Adverse Events (participants affected / at risk) | 116/513 | 113/518
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VVI 40 Pacing (N=513) | MVP Pacing (N=518)
Acute Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 6 (6) | 8 (8)
Cardiogenic Shock (General disorders) | 1 (1) | 2 (2)
Cerebellar Hematoma (General disorders) | 0 (0) | 1 (1)
Cerebral Hemorrhage (General disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chronic Obstructive Pulmonary Disorder with Renal Failure (General disorders) | 0 (0) | 1 (1)
Closed Head Trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 50 (91) | 53 (88)
Congestive Heart Failure with Acute Respiratory Distress Syndrome (General disorders) | 0 (0) | 1 (1)
Congestive Heart Failure with Anemia (General disorders) | 1 (1) | 0 (0)
Congestive Heart Failure with Angina (Cardiac disorders) | 1 (1) | 0 (0)
Congestive Heart Failure with Atrial Fibrillation (Cardiac disorders) | 2 (2) | 4 (4)
Congestive Heart Failure with Atrial Flutter (Cardiac disorders) | 1 (1) | 1 (1)
Congestive Heart Failure with Bronchitis (General disorders) | 1 (1) | 0 (0)
Congestive Heart Failure with Cellulitis and Anemia (General disorders) | 0 (0) | 1 (1)
Congestive Heart Failure with Chronic Obstructive Pulmonary Disease (General disorders) | 1 (1) | 0 (0)
Congestive Heart Failure with Coronary Artery Disease (General disorders) | 0 (0) | 1 (1)
Congestive Heart Failure with Coronary Artery Disease and Atrial Fibrillation (General disorders) | 0 (0) | 1 (1)
Congestive Heart Failure with Coronary Artery Disease, SVT and VT (General disorders) | 1 (1) | 0 (0) — Congestive Heart Failure with Coronary Artery Disease, Supraventricular Tachycardia (SVT) and Ventricular Tachycardia (VT)
Congestive Heart Failure with Infection - Respiratory Tract (General disorders) | 1 (1) | 0 (0)
Congestive Heart Failure with Myocardial Infarction (Cardiac disorders) | 2 (2) | 2 (2)
Congestive Heart Failure with Myocardial Infarction and Renal Failure (General disorders) | 0 (0) | 1 (1)
Congestive Heart Failure with Pneumonia (General disorders) | 2 (2) | 2 (2)
Congestive Heart Failure with Pneumonia and Renal Failure (General disorders) | 0 (0) | 1 (1)
Congestive Heart Failure with Pneumothorax and Right Atrial Lead Dislodgement (General disorders) | 0 (0) | 1 (1)
Congestive Heart Failure with Renal Failure (General disorders) | 0 (0) | 2 (2)
Congestive Heart Failure with Stroke (General disorders) | 1 (1) | 0 (0)
Congestive Heart Failure with Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Congestive Heart Failure with Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Coronary Artery Disease (Vascular disorders) | 3 (3) | 0 (0)
Coronary Artery Disease with Ventricular Tachycardia (General disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 3 (3) | 0 (0)
Hyperkalemia (General disorders) | 1 (1) | 1 (1)
Hypokalemia (General disorders) | 1 (1) | 0 (0)
Hypotension (General disorders) | 0 (0) | 2 (2)
Increased Right Ventricular Lead Impedance (General disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infection - Device, Leads (Infections and infestations) | 1 (1) | 4 (4)
Infection - Incision Site (Infections and infestations) | 0 (0) | 1 (1)
Infection - Pocket (Infections and infestations) | 2 (2) | 3 (3)
Infection - Systemic (Infections and infestations) | 1 (1) | 3 (3)
Infection - Urinary Tract (Infections and infestations) | 1 (1) | 1 (1)
Lead Dislodgement - Right Ventricular Lead (General disorders) | 0 (0) | 1 (1)
Lead Fracture - Right Ventricular Lead (General disorders) | 1 (1) | 3 (3)
Lead Perforation - Right Ventricular Lead (General disorders) | 0 (0) | 1 (1)
Lead Protrusion - Right Ventricular Lead (General disorders) | 0 (0) | 1 (1)
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukemia - Myelogenous (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Medication Allergy (General disorders) | 0 (0) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 16 (17) | 12 (13)
Myocardial Infarction with Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Necrosis - Left Lower Extremity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pantocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disease (Vascular disorders) | 2 (2) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural Effusion with Renal Failure and Sepsis (General disorders) | 0 (0) | 1 (1)
Pneumonia (General disorders) | 4 (4) | 2 (2)
Pneumonia with Myocardial Infarction (General disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Premature Battery Depletion (General disorders) | 0 (0) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary Embolus (General disorders) | 4 (4) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 6 (6) | 3 (4)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory Failure with Pneumonia and Atrial Fibrillation (General disorders) | 0 (0) | 1 (1)
Sepsis (General disorders) | 3 (5) | 3 (3)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stroke (General disorders) | 11 (12) | 5 (5)
Subdural Hematoma (General disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 11 (11) | 7 (8)
Ventricular Tachycardia and Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VVI 40 Pacing (N=513) | MVP Pacing (N=518)
Chest Pain (Cardiac disorders) | 36 (42) | 43 (51)
Congestive Heart Failure (Cardiac disorders) | 55 (73) | 44 (59)
Ventricular Tachycardia (Cardiac disorders) | 25 (30) | 26 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigational Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication.